CLINICAL TRIAL: NCT05383794
Title: Analysis of Gingival Crevicular Fluid Levels of miRNA 7a-5p, miRNA 21-3p, miRNA 21-5p, miRNA 200b-3p, miRNA 200b-5p, miRNA 100-5p, miRNA 125-5p in CVD and Periodontitis
Brief Title: Role of miRNAs in CVD and Periodontitis
Status: Completed | Type: Observational
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Other Study IDs: 215-21/PO
Record Dates: First submitted 2022-05-16; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Cardiovascular Diseases; Periodontal Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Evaluation of gingival crevicular fluid miRNA 7a-5p, miRNA 21-3p, miRNA 21-5p, miRNA 200b-3p, miRNA 200b-5p, miRNA 100-5p, miRNA 125-5p levels.
  Interventions: Other: Observation of Evaluation of gingival crevicular fluid miRNA 7a-5p, miRNA 21-3p, miRNA 21-5p, miRNA 200b-3p, miRNA 200b-5p, miRNA 100-5p, miRNA 125-5p levels.
- Periodontitis: Evaluation of gingival crevicular fluid miRNA 7a-5p, miRNA 21-3p, miRNA 21-5p, miRNA 200b-3p, miRNA 200b-5p, miRNA 100-5p, miRNA 125-5p levels.
  Interventions: Other: Observation of Evaluation of gingival crevicular fluid miRNA 7a-5p, miRNA 21-3p, miRNA 21-5p, miRNA 200b-3p, miRNA 200b-5p, miRNA 100-5p, miRNA 125-5p levels.
- Cardiovascular disease: Evaluation of gingival crevicular fluid miRNA 7a-5p, miRNA 21-3p, miRNA 21-5p, miRNA 200b-3p, miRNA 200b-5p, miRNA 100-5p, miRNA 125-5p levels.
  Interventions: Other: Observation of Evaluation of gingival crevicular fluid miRNA 7a-5p, miRNA 21-3p, miRNA 21-5p, miRNA 200b-3p, miRNA 200b-5p, miRNA 100-5p, miRNA 125-5p levels.
- Periodontitis + cardiovascular disease: Evaluation of gingival crevicular fluid miRNA 7a-5p, miRNA 21-3p, miRNA 21-5p, miRNA 200b-3p, miRNA 200b-5p, miRNA 100-5p, miRNA 125-5p levels.
  Interventions: Other: Observation of Evaluation of gingival crevicular fluid miRNA 7a-5p, miRNA 21-3p, miRNA 21-5p, miRNA 200b-3p, miRNA 200b-5p, miRNA 100-5p, miRNA 125-5p levels.

INTERVENTIONS:
Other: Observation of Evaluation of gingival crevicular fluid miRNA 7a-5p, miRNA 21-3p, miRNA 21-5p, miRNA 200b-3p, miRNA 200b-5p, miRNA 100-5p, miRNA 125-5p levels. — Evaluation of gingival crevicular fluid miRNA 7a-5p, miRNA 21-3p, miRNA 21-5p, miRNA 200b-3p, miRNA 200b-5p, miRNA 100-5p, miRNA 125-5p levels.

SUMMARY:
Several micro-RNA plays a key role in endothelial function and may be a link for the known interaction of periodontitis and cardiovascular disease. The investigators compared the impact of gingival health, periodontitis (CP), cardiovascular disease or of both diseases (CP +cardiovascular disease) on gingival crevicular fluid miRNA 7a-5p, miRNA 21-3p, miRNA 21-5p, miRNA 200b-3p, miRNA 200b-5p, miRNA 100-5p, miRNA 125-5p levels.

DETAILED DESCRIPTION:
The investigators compared the impact of gingival health, periodontitis (CP), cardiovascular disease or of both diseases (CP +cardiovascular disease) on gingival crevicular fluid miRNA 7a-5p, miRNA 21-3p, miRNA 21-5p, miRNA 200b-3p, miRNA 200b-5p, miRNA 100-5p, miRNA 125-5p levels.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 15 teeth
* CP with a minimum of 40% of sites with a clinical attachment level (CAL)

  ≥2mm and probing depth (PD) ≥4mm;
* Presence of at least ≥2 mm of crestal alveolar bone loss verified on digital periapical radiographs
* Presence of ≥40% sites with bleeding on probing (BOP)

Exclusion Criteria:

* Intake of contraceptives
* Intake of immunosuppressive or anti-inflammatory drugs throughout the last three months prior to the study
* Status of pregnancy or lactation
* Previous history of excessive drinking
* Allergy to local anaesthetic
* Intake of drugs that may potentially determine gingival hyperplasia such as Hydantoin, Nifedipine, Cyclosporin A or similar drugs.

Age Groups: Child, Adult, Older Adult
Study Population: healthy controls (n=28), periodontitis (n=30), CVD (n=28), and a combination of periodontitis + CVD (n=29)
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment level | 1-year
  Evaluation of changes (in millimeters) of Clinical attachment level loss

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — Università degli Studi di Catania
Locations (1):
- University of Catania, Catania, CT, Italy

IPD SHARING:
Plan to Share IPD: Undecided
all collected IPD, all IPD that underlie results in a publication